CLINICAL TRIAL: NCT01411930
Title: Acute Impact of IM Aripiprazole and Olanzapine on Insulin Resistance in High Risk Prediabetics
Brief Title: Acute Impact of Intramuscular (IM) Aripiprazole and Olanzapine on Insulin Resistance in High Risk Prediabetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jonathan M. Meyer, MD, Research Scientist, Veterans Medical Research Foundation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 080225
Record Dates: First submitted 2009-09-15; First posted 2011-08-08 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes
Keywords: Insulin resistance; Antipsychotics; Olanzapine; Aripiprazole
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Aripiprazole; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine -> Aripiprazole (Experimental): Crossover design. Order of agents is randomized. For this arm, the order will be IM olanzapine (1st clamp study) and IM aripiprazole (2nd clamp study).
  Interventions: Drug: Intramuscular olanzapine, aripiprazole
- Aripiprazole -> Olanzapine (Experimental): Crossover design. Order of agents is randomized. For this arm, the order will be IM aripiprazole (1st clamp study) and IM olanzapine (2nd clamp study).
  Interventions: Drug: Intramuscular aripiprazole, olanzapine

INTERVENTIONS:
Drug: Intramuscular olanzapine, aripiprazole — 1. 1st clamp: single intramuscular 10.0 mg dose of olanzapine
  2. 2nd clamp: single intramuscular 9.75 mg dose of aripiprazole
  Other Names: Olanzapine -> Aripiprazole
  Arms: Olanzapine -> Aripiprazole
Drug: Intramuscular aripiprazole, olanzapine — 1. 1st clamp: single intramuscular 9.75 mg dose of aripiprazole
  2. 2nd clamp: single intramuscular 10.0 mg dose of olanzapine
  Other Names: Aripiprazole -> Olanzapine
  Arms: Aripiprazole -> Olanzapine

SUMMARY:
Antipsychotic medicines used to treat mental illnesses have been associated with effects on blood sugar control. Laboratory studies have shown that certain medications in particular may alter how insulin works. One purpose of this study is determine if antipsychotic medications have immediate effects on insulin action in individuals who do not have a mental disorder, but who have risk factors for diabetes. A second purpose is to demonstrate the feasibility of using volunteers without psychiatric disorders, and who do not take psychiatric medications, as a means for studying antipsychotic metabolic effects.

DETAILED DESCRIPTION:
Antipsychotic medications are those that treat the most severe psychiatric symptoms, such as hallucinations, paranoid thoughts, and delusions. Research shows that some of these medications may put people at a higher risk of metabolic derangements, such as insulin resistance. Certain antipsychotics, like clozapine and olanzapine, are associated with a higher risk of metabolic side effects than others, like aripiprazole and ziprasidone. This study will compare the effects of single doses of two antipsychotic medications, olanzapine and aripiprazole, on insulin action in nonpsychiatrically ill volunteer subjects.

Participation in this study will last 6 weeks. Participants will first complete a screening visit that will include the following: an oral glucose tolerance test (OGTT), which involves a blood draw, consumption of a sugar drink, and then a second blood draw; a review of medical and psychiatric history, including use of medicines and psychiatric medications; and measurement of participants' height and weight. The second visit, scheduled 2 weeks after screening, will include a tracer-clamp study to test how participants' bodies handle sugar. The tracer-clamp study will be conducted over the course of one night and morning and will require participants to stay at the study location overnight. At 3 AM, participants will receive an intravenous line (IV) with a sugar solution. Just before 8 AM, they will receive a second IV in the opposite arm that will draw blood and monitor blood sugar levels.

At 8 AM, participants will begin receiving insulin in the first IV; blood samples will be drawn and blood sugar levels will be monitored during this time to ensure they remain within a healthy range. At 11 AM, participants will receive an injection of an antipsychotic medication into their arm muscles. The antipsychotic, which will be randomly assigned, will be either olanzapine or aripiprazole. Participants will be monitored for 3 hours after receiving the injection of antipsychotic medication; during this time, more blood samples will be drawn, blood sugar levels will be monitored to ensure they are within a healthy range, and secondary medications will be available to counteract certain side effects of the antipsychotics.

After 4 more weeks, participants will undergo a 2nd tracer-clamp study, this time receiving the antipsychotic not given in the first clamp study. The protocol for this visit is otherwise identical to the first clamp study.

ELIGIBILITY:
Inclusion Criteria:

* No history of axis I mood, anxiety or psychotic disorder (confirmed by Structured Clinical Interview for DSM-IV), and taking no psychotropics
* Prediabetic, based on a finding of impaired glucose tolerance (2 hour post-load serum glucose 140-199 mg/dl) on a 75 gram standard oral glucose tolerance test within the past 90 days
* Family history of type 2 diabetes mellitus
* BMI 25-35 kg/m2
* Males, ages 40-65 inclusive
* English speaker with ability to provide informed consent
* Nonsmoker

Exclusion Criteria:

* History of Axis I Mood, Anxiety or Psychotic Disorder or Use of Psychotropics

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 6 weeks
  2 overnight procedures 4 weeks apart, plus screening procedure

SECONDARY OUTCOMES:
Hepatic glucose production | 6 weeks
  2 overnight procedures 4 weeks apart, plus screening procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Meyer, MD, Principal Investigator — VA San Diego and VMRF
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States